CLINICAL TRIAL: NCT02882269
Title: A Randomized Controlled Clinical Trial to Investigate the Effect of Neoadjuvant Chemotherapy for the Treatment of Resectable Locally Advanced Colon Cancer
Brief Title: Neoadjuvant Chemotherapy for the Treatment of Resectable Locally Advanced Colon Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRSYM201608
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Colon Cancer
Keywords: locally advanced colon cancer; neoadjuvant chemotherapy
MeSH Terms: conditions — Colonic Neoplasms | interventions — Drug Combinations; Folfox protocol; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Postoperative chemotherapy (Active Comparator): Patients receive 6 months of chemotherapy after surgery.
  Interventions: Drug: Postoperative chemotherapy
- Neoadjuvant chemotherapy (Experimental): Patients receive 3-4 cycles of chemotherapy before surgery. Preoperative and postoperative chemotherapy will be given for a total of 6 months.
  Interventions: Drug: Neoadjuvant chemotherapy

INTERVENTIONS:
Drug: Postoperative chemotherapy — Locally advanced colon cancer patients will receive surgery first, followed by 6 months of chemotherapy. The recommended chemotherapy regimes includes FOLFOX, CapeOX, FOLFIRI, Capecitabine monotherapy.
  Other Names: drug combination (FOLFOX, CapeOX or FOLFIRI) or Capecitabine monotherapy
  Arms: Postoperative chemotherapy
Drug: Neoadjuvant chemotherapy — Neoadjuvant chemotherapy will be given to locally advanced colon cancer patients for 3-4 cycles. Surgery will be performed between 3 to 4 weeks subsequent to the last cycle of chemotherapy. After surgery, additional chemotherapy will be given. Preoperative and postoperative chemotherapy will be given for a total of 6 months. The recommended chemotherapy regimes includes FOLFOX, CapeOX, FOLFIRI, Capecitabine monotherapy.
  Other Names: drug combination (FOLFOX, CapeOX or FOLFIRI) or Capecitabine monotherapy
  Arms: Neoadjuvant chemotherapy

SUMMARY:
A randomized controlled clinical trial to compare the short and long outcomes of Neoadjuvant chemotherapy with postoperative chemotherapy in patients with resectable locally advanced colon cancer

DETAILED DESCRIPTION:
For resectable locally advanced colon cancer, the preferred treatment is colectomy with en bloc removal of the regional lymph nodes followed by chemotherapy of about 6 months. However, surgery may postpone the administration of chemotherapy due to postoperative complications such as anastomosis leakage, abdominal infection, thus leads to a poor survival. Some scholars suggested that for patients with locally advanced colon cancer, chemotherapy given before surgery might shrink or downstage tumor, facilitate surgery and promote a better oncological outcome. Whether adjuvant chemotherapy benefits these patients with better outcome still remains controversial.

In this study, eligible patients will be randomly allocated to receive either adjuvant chemotherapy or not. For patients receiving adjuvant chemotherapy, surgery will be performed 3-4 weeks later. Preoperative and postoperative chemotherapy will be given for a total of about 6 months. For patients receiving no preoperative chemotherapy, chemotherapy will be given for about 6 months postoperatively. The recommended chemotherapy regimes includes FOLFOX, CapeOX, FOLFIRI, Capecitabine monotherapy. Patients will be followed up every 3 months for 2 year, every 6 months for 3 years postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients suitable for curative surgery between 18 to 80 years old;
* American Society of Anesthesiologists(ASA) grade I-III;
* Pathological diagnosis of adenocarcinoma;
* Tumor located between the cecum and sigmoid colon;
* Enhanced CT scan of chest, abdominal and pelvic cavity: preoperative assessment of tumor stage is T3-T4 N0 or T any N+ (according to the National Comprehensive Cancer Network(NCCN) clinical practice guidelines in oncology: colon cancer version 2.2015);there is no distant metastasis;
* Informed consent;
* No preoperative chemoradiotherapy;
* No history of familial adenomatous polyposis, ulcerative colitis or Crohn's disease.

Exclusion Criteria:

* Pregnant patient;
* History of psychiatric disease;
* Use of systemic steroids;
* Simultaneous multiple primary colorectal cancer;
* Preoperative imaging examination results show:

  1. distant metastasis;
  2. unable to perform R0 resection;
* Postoperative pathology of T1-T2 N0;
* History of any other malignant tumor in recent 5 years;
* Patients need emergency operation: mechanic ileus, perforation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-12; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 3 years

SECONDARY OUTCOMES:
overall survival | 3 years
recurrence-free survival | 3 years
local recurrence rate | 3 years
length of postoperative hospital stay | 30 days
  Length of postoperative hospital stay is defined as a duration between surgery and first discharge. An expected average is 10 days.
early complication rate | 30 days
  Early complication is defined as a complication that occurred between the finish of the surgery and postoperative day 30. Complications includes anastomotic leakage, anastomotic bleeding, chyle leakage, wound infection, pulmonary embolism, myocardial infarction et al.The Clavien-Dindo Classification of Surgical Complications will be applied to access the degree of severity of postoperative complications.
operative time | 1 day
number of lymph nodes retrieved | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Fumin Zhang, Professor, Study Director — Ethics Committee of the First Affiliated Hospital, Nanjing Medical University, Jiangsu Province Hospital

IPD SHARING:
Plan to Share IPD: No